CLINICAL TRIAL: NCT01667484
Title: Does Adderall XR Improve Processing Speed in Cognitively Impaired MS Patients?
Brief Title: Adderall XR and Processing Speed in Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Sarah Morrow, Assistant Professor of Neurology, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102774
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Impaired Processing Speed; Cognitive Impairment; Multiple Sclerosis
Keywords: Cognitive Impairment; Multiple Sclerosis; Processing Speed; Treatment
MeSH Terms: conditions — Cognitive Dysfunction; Multiple Sclerosis | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): treatment group #1
  Interventions: Drug: Placebo
- Adderall XR 5mg (Active Comparator): treatment group #2
  Interventions: Drug: Adderall XR 5mg
- Adderal XR 10mg (Active Comparator): treatment group #3
  Interventions: Drug: Adderall XR 10 mg

INTERVENTIONS:
Drug: Adderall XR 5mg
  Arms: Adderall XR 5mg
Drug: Adderall XR 10 mg
  Arms: Adderal XR 10mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Cognitive impairment, or problems with thinking and memory, is common in multiple sclerosis (MS) and can occur independently of physical disability. It is the most common reason, along with physical fatigue, for MS patients to stop working. The most frequent complaint is problems with multi-tasking or thinking quickly, which corresponds to impairment in the cognitive domain of processing speed. Currently there is treatment available to prevent relapses and physical disability but there are no medications that have been shown to treat cognitive impairment. Amphetamines have been beneficial for selective attention and processing speed in attention deficit hyperactivity disorder (ADHD) and traumatic brain injury. This is study will determine whether Adderall XR improves objective measures of processing speed and attention in MS patients impaired in this cognitive domain, by comparing two doses of Adderall XR (5 and 10mg) to placebo before and after the medication is administered. The results of this study will help provide data to design a larger study to determine if Adderall XR, and potentially other amphetamine drugs, will help treat cognitive impairment in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* - Males/Females who are ≥ 18 years old and ≤ 59 years old
* Relapsing Remitting, Secondary Progressive or Primary Progressive MS, as per revised McDonald's Criteria
* Have not received corticosteroids in last thirty days or a relapse in the last ninety days
* An Expanded Disability Status Scale (EDSS) of ≤ 6.5
* If female, must neither be pregnant nor breast-feeding

Exclusion Criteria:

* - Have evidence of other medical cause(s) of cognitive impairment
* Have evidence of major depression as determined by a positive Beck Depression Index-Fast screen ≥ 13and/or by clinician interview or evidence of severe fatigue with a Fatigue Severity Scale ≥ 5.
* Have demonstrated a hypersensitivity to amphetamines in the past
* Have uncontrolled or labile hypertension (> 135/85 mm Hg, treated or untreated)
* Have a history of structural heart disease, including atherosclerosis or angina
* Have a diagnosis of bipolar disorder or a history of a psychotic episode
* The following medications are not permitted to be used within 14 days the study

  1. Monoamine Oxidase Inhibitors
  2. Sympathomimetics or methadone
  3. Antipsychotic agents
  4. Modafinil
* The following medications are permitted if the dose has been stable for ≥ 28 days

  1. Short acting benzodiazepines, qhs administration only
  2. Anticonvulsants, including gabapentin and pregabalin
  3. Bupropion
  4. Tricyclic Antidepressants
  5. Anti-spasmodics such as baclofen or tizanidine
  6. Anticholinergic medication
  7. Selective serotonin(-norepinephrine) reuptake inhibitors

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in score of Paced Auditory Serial Addition Test (PASAT) | pre and 7 hours post dose
  measure of processing speed
Change in Score of Symbol Digit Modalities Test (SDMT) | pre and 7 hours post dose
  measure of processing speed

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Morrow, MD, MS, FRCPC, Principal Investigator — London Health Sciences Center
Locations (1):
- London Health Sciences Center and St. Joseph's Heathcare Center (Parkwood), London, Ontario, Canada